CLINICAL TRIAL: NCT03914352
Title: A Novel Immunotherapy PD-1 Antiboty to Suppress Recurrence of Hepatocellular Carcinoma Combined With Portal Vein Thrombus After Hepatic Resection
Brief Title: A Novel Immunotherapy PD-1 Antiboty to Suppress Recurrence of HCC Combined With PVTT After Hepatic Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jia-zhou Ye, Principal investigator, Cancer Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHGuangxiMU
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Portal vein tumor thrombus; Hepatic resection; Recurrence; PD-1 antibody
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — spartalizumab; camrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PD-1 antibody group (Experimental): In this group participants were treated with PD-1 antibody (240mg, Intravenous drip infusion, Q14 days) since the15 days after hepatic resection and at the interval of 15 days.
  Interventions: Drug: PD-1 antibody
- Controlled group (Active Comparator): In this group entrolled patients were treated with TACE in the 30 days after hepatic resection.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: PD-1 antibody — In this group participants were treated with PD-1 antibody (240mg, Intravenous drip infusion, Q14 days) since the15 days after hepatic resection and at the interval of 15 days.
  Other Names: SHR-1210
  Arms: PD-1 antibody group
Procedure: TACE — In this group enrolled patients were treated with TACE at the30 days after hepatic resection.
  Arms: Controlled group

SUMMARY:
Hepatic resection is the most effective curative treatment for resectable HCC, whereas frequent recurrence usually impaired the efficacy of hepatic resection and contributed poor survivals. PVTT has been certified as an independent risk of early recurrence.

Although TACE has been used to decrease the intraheptic recurrence. However, the intraheptic recurrence rate remains high and meanwhile it is uncapable to suppress extrahepatic recurrence. In addition, systematic therapy the small molecular target antiangiogenesis medicine sorafenib were used to prevent recurrence. Unfortunately, the STORM trial shows that postoperative antiangiogenesis therapy was failed to suppress recurrence and prolong survival period for HCC patients. Thus, novel effective systematic therapy to suppress postoperative recurrence is in urgent need.

At present, the PD-1 antibody has presented a promising and safe therapeutic result of unresectable HCC and provided good survival benefit for advanced HCC patients. Consistent with this, we proposed a hypothesis that a novel immunetherapy using the PD-1 antibody could suppress postoperative recurrence and prolong HCC patients survival period effectively.

DETAILED DESCRIPTION:
Hepatic resection is the most effective curative treatment for resectable hepatocellular carcinoma (HCC), whereas frequent recurrence usually impaired the efficacy of hepatic resection and contributed poor survivals. Portal vein tumor thrombus (PVTT) has been certified as an independent risk of early recurrence (≤2years after hepatic resection).

Although Transarterial Chemoembolization (TACE) has been used as an effective local adjuvant treatment to decrease the intraheptic recurrence. However, the intraheptic recurrence rate remains high and meanwhile it is uncapable to suppress extrahepatic recurrence. In addition, systematic therapy the small molecular target antiangiogenesis medicine sorafenib were used to prevent recurrence. Unfortunately, the double blind randomized STORM trial shows a negative result that postoperative antiangiogenesis therapy was failed to suppress recurrence and prolong survival period for HCC patients. Thus, novel effective systematic therapy to suppress postoperative recurrence is in urgent need.

At present, the PD-1 antibody has presented a promising and safe therapeutic result of unresectable HCC and provided good survival benefit for advanced HCC patients. Consistent with this, we proposed a hypothesis that a novel immunetherapy using the PD-1 antibody could suppress postoperative recurrence and prolong HCC patients survival period effectively.

ELIGIBILITY:
Inclusion Criteria:

* HCC comfirmed by postoperative histology examination
* PVTT comfirmed by postoperative histology examination
* None other type of malignant tumors
* None intra or extra-hepatic recurrence postoperative adjuvant therapy
* Child-pugh grade A or B liver function
* None other organ dysfunction

Exclusion Criteria:

* Combined with other type of malignant tumors
* Presence of intra or extra-hepatic recurrence
* Child-pugh grade C liver function
* Combined with other organ dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Cumulative survival period after hepatic resection
Disease-free survival | 5 years
  Cumulative none recurrence survival period after hepatic resection

CONTACTS AND LOCATIONS:
Overall Officials: Lequn Li, M.D., Study Chair — Cancer Hospital of Guangxi Medical University; Jiazhou Ye, M.D., Principal Investigator — Cancer Hospital of Guangxi Medical University
Locations (1):
- Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No